CLINICAL TRIAL: NCT03857958
Title: Comparison of Metal Versus Plastic Side-by-side Stent Insertion in Malignant Hilar Biliary Obstruction
Brief Title: Metal Versus Plastic Stent in Malignant Hilar Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1812-098-996
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Malignant Hepatobiliary Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCSEMS (Experimental): In patients with malignant hilar biliary obstruction, endoscopic drainage is performed for biliary drainage. Since intrahepatic bile ducts are separated, it is preferable to insert a stent into bilateral intrahepatic bile ducts for bile drainage if possible. In FCSEMS group, patients are inserted with Fully covered self-expandable metal stent (FCSEMS) bilaterally for malignant hilar biliary stricture via endoscopic retrograde cholangio-pancreatography.
  Interventions: Procedure: endoscopic retrograde cholangio-pancreatography
- Plastic stent (Active Comparator): In patients with malignant hilar biliary obstruction, endoscopic drainage is performed for biliary drainage. Since intrahepatic bile ducts are separated, it is preferable to insert a stent into bilateral intrahepatic bile ducts for bile drainage if possible. In plastic stent group, patients are inserted with plastic stents bilaterally for malignant hilar biliary stricture.
  Interventions: Procedure: endoscopic retrograde cholangio-pancreatography

INTERVENTIONS:
Procedure: endoscopic retrograde cholangio-pancreatography — In patients who were identified to have malignant hilar biliary obstruction, bilateral stents insertion is attempted via ERCP. There will be two groups divided by stent material; FCSEMS and Plastic stent.
  Other Names: Plastic stent; FCSEMS

SUMMARY:
The purpose of this study was to compare the difference in the stent patency duration between side-by-side fully covered self-expanding metal stents (SEMS) and side-by-side plastic stents in patients with malignant hilar biliary obstruction.

DETAILED DESCRIPTION:
In the case of distal common bile duct obstruction, the SEMS was reported to be clinically superior to the plastic stent in previous studies. However, there are few studies comparing the two methods in patients with malignant hilar biliary obstruction. In contrast to the distal common bile duct obstruction, the advantage of plastic stents over SEMSs exists, and plastic stents are used commonly in real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable malignant hilar biliary stricture requiring biliary drainage through endoscopic procedure

Exclusion Criteria:

* If endoscopy is not possible based on the judgement of the researcher
* Life expectancy less than 6 months
* Acute cholecystitis
* Previous history of percutaneous transhepatic biliary drainage
* Previous history of metal stent placement for malignant biliary stricture

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of stent patency | 9 months after randomization.
  The period from the insertion of the stent to the point at which stent revision is required.

CONTACTS AND LOCATIONS:
Overall Officials: Seoul National University Hospital Seoul National University Hospital, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea